CLINICAL TRIAL: NCT07401472
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered BW-50218 in Healthy Participants
Brief Title: Phase 1, Single Ascending Dose Study of BW-50218 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Argo Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BW-50218-1001
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants Study
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- BW-50218 Dose 1 (Experimental): Single dose of BW-50218 injection (Dose 1).
  Interventions: Drug: BW-50218 Injection
- BW-50218 Dose 2 (Experimental): Single dose of BW-50218 injection (Dose 2).
  Interventions: Drug: BW-50218 Injection
- BW-50218 Dose 3 (Experimental): Single dose of BW-50218 injection (Dose 3).
  Interventions: Drug: BW-50218 Injection
- BW-50218 Dose 4 (Experimental): Single dose of BW-50218 injection (Dose 4).
  Interventions: Drug: BW-50218 Injection
- BW-50218 Dose 5 (Experimental): Single dose of BW-50218 injection (Dose 5).
  Interventions: Drug: BW-50218 Injection
- BW-50218 Dose 6 (Experimental): Single dose of BW-50218 injection (Dose 6).
  Interventions: Drug: BW-50218 Injection
- Saline Placebo (Placebo Comparator): Single dose of Saline Placebo
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Drug: BW-50218 Injection — Solution for injection
  Arms: BW-50218 Dose 1; BW-50218 Dose 2; BW-50218 Dose 3; BW-50218 Dose 4; BW-50218 Dose 5; BW-50218 Dose 6
Drug: Saline (0.9% NaCl) — Solution for injection
  Arms: Saline Placebo

SUMMARY:
Phase 1, Single Ascending Dose Study of Subcutaneous BW-50218 in Healthy Participants

DETAILED DESCRIPTION:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered BW-50218 in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing written informed consent and complying with all study procedures for the duration of the study.
* Body weight and body mass index (BMI) within a range considered appropriate for study participation by the investigator.
* Female participants must be non-pregnant, non-lactating, and either of non-childbearing potential or using highly effective contraception.
* Male participants with partners of childbearing potential must agree to use effective contraception.

Exclusion Criteria:

* Any medical condition, recent illness, or laboratory result that, in the investigator's opinion, may increase risk or interfere with participation in the study.
* Recent hospitalization or a significant acute medical event.
* History of cancer or any long-term medical condition that the study doctor considers clinically relevant.
* Clinical laboratory findings outside of range which are deemed clinically significant by the investigator at screening or Day -1.
* Positive test for hepatitis B, hepatitis C, or HIV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From baseline up to Day 360 (End of Study)
  Evaluation of the number of participants with treatment-emergent adverse events and serious adverse events. The severity of AEs will be assessed and categorized according to the "Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" (FDA, 2007).
Change from Baseline in Clinical Laboratory Test Results | From baseline up to Day 360 (End of Study)
  Evaluation of hematology, clinical chemistry, and urinalysis parameters.
Change from Baseline in Vital Signs | From baseline up to Day 360 (End of Study)
  Evaluation of blood pressure, heart rate, respiratory rate, and body temperature.
Change from Baseline in 12-Lead Electrocardiogram (ECG) Parameters | From baseline up to Day 360 (End of Study)
  Evaluation of PR, QRS, QT, and QTc intervals.
Change from Baseline in Physical Examination Findings | From baseline up to Day 360 (End of Study)
  Assessment of clinically significant changes in physical examination findings.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | From pre-dose up to Day 8
  Evaluation of the maximum plasma concentration of BW-50218.
Time to Maximum Plasma Concentration (Tmax) | From pre-dose up to Day 8
  Evaluation of the time to reach maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve (AUC) | From pre-dose up to Day 8
  Evaluation of AUC from time zero to 24 hours (AUC0-24), to 48 hours (AUC0-48), and to infinity (AUC0-inf).
Terminal Elimination Half-Life (t1/2) | From pre-dose up to Day 8
  Evaluation of the elimination half-life of BW-50218.
Urine Pharmacokinetic Parameters | From pre-dose up to 24 hours post-dose
  Evaluation of urine output (Aet) and renal clearance (CLr).
Change from Baseline in Serum Transthyretin (TTR) Protein Concentration | From baseline up to Day 360 (End of Study)
  Assessment of the concentration of Transthyretin (TTR) protein in serum to evaluate pharmacodynamic response.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqiong Li, MD, Study Director — Shanghai Argo Biopharmaceutical Co., Ltd.

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding sharing of de-identified IPD will be made by the Sponsor after study completion and will consider scientific merit, participant privacy, and regulatory requirements.